CLINICAL TRIAL: NCT04678557
Title: An Open-Label Phase 1/2 Study to Evaluate the Safety, Engraftment, and Efficacy of VC-01™Combination Product in Subjects With Type 1 Diabetes Mellitus [T1DM]
Brief Title: A Study to Evaluate Safety, Engraftment, and Efficacy of VC-01 in Subjects With T1 Diabetes Mellitus
Acronym: VC01-103
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient functional product engraftment
Sponsor: ViaCyte (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: VC01-103
Record Dates: First submitted 2020-11-30; First posted 2020-12-22 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: There are two Cohorts in this study design. Cohort 1 (Phase 1) enrolls up to 30 subjects total. After Cohort 1 enrollment is completed, Cohort 2 enrollment then occurs with up to an additional 40 subjects. A total of up to 70 subjects will be enrolled under this Phase 1/2 protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sentinel units (aka Cohort 1) (Experimental): VC-01 Combination Product; Up to ten (10) VC-01 sentinels
  Interventions: Combination Product: VC-01 Combination Product
- Dose-finding units (aka Cohort 2) (Experimental): VC-01 Combination Product; Up to twelve units implanted of which up to nine (9) are VC-01-DF (dose-finding) implants and the rest are VC-01 sentinels
  Interventions: Combination Product: VC-01 Combination Product

INTERVENTIONS:
Combination Product: VC-01 Combination Product — PEC-01 cells loaded into an Encaptra Drug Delivery System
  Other Names: PEC-Encap

SUMMARY:
VC01-103 will evaluate an experimental combination product, cell replacement therapy intended to provide a functional cure to subjects with Type 1 Diabetes.

DETAILED DESCRIPTION:
This trial will test if VC-01 combination product can be implanted and maintained with safety, tolerability, and efficacy for up to Month 12/Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant women
* Diagnosis of T1DM for a minimum of 3 years.
* Stable, optimized diabetic regimen
* Acceptable candidate for implant and explant procedures.
* Willing and able to comply with protocol requirements.
* Meet insulin dosing requirements per protocol

Exclusion Criteria:

• Advanced complications associated with diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manasi Jaiman, MD, Principal Investigator — ViaCyte, Inc.
Locations (4):
- United States (4):
  - AMCR Institute, Escondido, California
  - Diablo Clinical Research, Walnut Creek, California
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Texas Diabetes & Endocrinology, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 8 or 10 Sentinel Units Implanted (Cohort 1): VC-01 combination product is comprised of PEC-01 cells loaded into an Encaptra Drug Delivery System. In Cohort 1 of this study, 8 or 10 VC-01 sentinel units were surgically implanted in each subject during a single procedure. Sentinel units are smaller versions of the product not intended to provide efficacy but are instead explanted at various timepoints over the course of the study and examined histologically.
- 9 Dose Finding Units Implanted (Cohort 2): A total of 12 VC-01 units were implanted in each of the Cohort 2 subjects in a single surgical procedure. Of those units, 9 were VC-01 Dose Finding (DF) units. DF units are larger than sentinels and intended to remain implanted during the duration of participation in the trial to assess efficacy.
  The remaining 3 units implanted were the smaller VC-01 sentinel units intended for explant at various time points for analysis histologically.
Period: Overall Study
Arm/Group | 8 or 10 Sentinel Units Implanted (Cohort 1) | 9 Dose Finding Units Implanted (Cohort 2)
Started | 17 | 14
Completed | 16 | 0
Not Completed | 1 | 14
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lack of Efficacy | 0 | 13
Not completed — Safety Evaluation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sentinel Units (Aka Cohort 1) | Dose-finding Units (Aka Cohort 2) | Total
Number analyzed (Participants) | 17 | 14 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (13.11) | 44.1 (8.53) | 40.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 14 | 31
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.98 (2.992) | 27.28 (2.807) | 26.00 (3.09)
Duration of Type 1 Diabetes [Mean (Standard Deviation); unit: years] | 19.4 (12.08) | 26.4 (11.24) | 22.5 (12.0)

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: The Percentage of Graft Cells Present at Post-implant Time Points Relative to Pre-clinical Models
Description: Through histology, the potential for functional engraftment of VC-01 combination product could be assessed in Cohort 1 subjects. Explanted sentinel units from subjects were processed and stained for markers identifying the number of graft cell nuclei (i.e., signifying the cells were viable). The percentage of viable graft cells in these explanted units were then compared to the percentage of viable graft cells from the pre-clinical (i.e., animal) models. These pre-clinical models are based on animal studies performed at ViaCyte (ref: internal study report). The data in Outcome Measure Data Table represent the % of viable graft cells present in the explanted sentinels compared to what was expected based on the animal model at Weeks 4, 8, 12, and 26 (e.g., At Week 4, there was an average of 18.27% viable graft cells in the participant's explants compared to what was expected based on the animal models).
Time Frame: Weeks 4, 8, 12 and 26
Population: For each timepoint, explanted sentinel units containing PEC-01 cells from the 17 subjects were stained and evaluated for graft cell survival (i.e., viability). Not all subjects had units explanted at every timepoint, and units explanted that had "de minimus" graft cell survival (i.e., minimal, < 500 cells, < 4% of pre-clinical controls) could not be evaluated and were not included in the summary table.
Measure: Mean (Standard Deviation); unit: %cells in sentinels rel to animal models
Units Other Than Participants: VC01 sentinels (contains PEC-01 cells)
Arm/Group | Sentinel Units (Aka Cohort 1)
Number analyzed (Participants) | 17
Number analyzed (VC01 sentinels (contains PEC-01 cells)) | 81
%cells in sentinels rel to animal models
  Week 4: number analyzed (Participants) | 10
  Week 4: number analyzed (VC01 sentinels (contains PEC-01 cells)) | 45
  Week 4 | 18.27 (13.94)
  Week 8: number analyzed (Participants) | 5
  Week 8: number analyzed (VC01 sentinels (contains PEC-01 cells)) | 8
  Week 8 | 6.23 (4.63)
  Week 12: number analyzed (Participants) | 11
  Week 12: number analyzed (VC01 sentinels (contains PEC-01 cells)) | 23
  Week 12 | 7.58 (7.27)
  Week 26: number analyzed (Participants) | 3
  Week 26: number analyzed (VC01 sentinels (contains PEC-01 cells)) | 5
  Week 26 | 8.02 (8.09)

2. Primary Outcome: Cohort 2: The Change in AUC (Area Under Curve) From Baseline to Week 26 in C-peptide During 4-hour MMTT
Description: Evaluation of clinical efficacy of VC-01 combination product in Cohort 2 subjects was intended by measuring C-peptide levels during a 4-hour Mixed Meal Tolerance Test (MMTT). Blood glucose and C-peptide data were collected from subjects at timepoints 0, 30, 60, 90, 120, 180, 240 minutes after ingestion of a "meal" (i.e., BOOST drink). These C-peptide data points could be used to create the AUC calculation. If the implanted units contained mature, insulin-producing cells, stimulated C-peptide levels would be expected to increase over the time course in reaction to the meal.
Time Frame: To Week 26
Population: Stimulated C-peptide data from the MMTT showed every value from baseline and Week 26 samples at all timepoints to be "undetectable" (<0.1 ng/mL) except for one subject for whom the AUC could be calculated. Analyzing the data was deemed futile because the number of surviving graft cells was noted as insufficient for establishing the biological critical mass. The change from baseline to Week 26 in AUC for this one subject is provided below.
Measure: Number; unit: ng*h/mL
Arm/Group | Dose-finding Units (Aka Cohort 2)
Number analyzed (Participants) | 1
ng*h/mL | 0.325

ADVERSE EVENTS:
Time Frame: Cohort 1 subjects reported adverse events over approximately 7 months (e.g., subjects implanted/treated for 6 months). Cohort 2 subjects reported adverse events over approximately 13 months (e.g., subjects implanted/treated for 12 months).
Description: AE/SAE Definitions used are the same as the ClinicalTrials.gov definitions.
  Systematic Assessment of AE Collection was used (e.g., regular investigator assessment was required at each study visit per protocol). In addition, routine monitoring visits to the site provided 100% source document verification of the AE Collection.
Arm/Group | Sentinel Units (Aka Cohort 1) | Dose-finding Units (Aka Cohort 2)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/17 | 3/14
Other Adverse Events (participants affected / at risk) | 17/17 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sentinel Units (Aka Cohort 1) (N=17) | Dose-finding Units (Aka Cohort 2) (N=14)
Vanishing Twin Syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Subarachnoid hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sentinel Units (Aka Cohort 1) (N=17) | Dose-finding Units (Aka Cohort 2) (N=14)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 6 (7)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5) | 3 (6)
Vomiting (Gastrointestinal disorders) | 4 (5) | 2 (2)
Complication of Device Removal (General disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
Implant Site Erythema (General disorders) | 0 (0) | 2 (5)
Implant Site Hypoaesthesia (General disorders) | 2 (2) | 0 (0)
Infusion Site Haemorrhage (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Postoperative wound infection (Infections and infestations) | 2 (2) | 1 (2)
Incision site complication (Injury, poisoning and procedural complications) | 3 (3) | 3 (6)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1) | 1 (3)
Incision site haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Incision site hypoaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Incision site pain (Injury, poisoning and procedural complications) | 15 (30) | 12 (60)
Incision site pruritis (Injury, poisoning and procedural complications) | 1 (1) | 1 (6)
Incision site rash (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision site swelling (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Post procedural contusion (Injury, poisoning and procedural complications) | 1 (1) | 7 (12)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (2) | 5 (6)
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 4 (8)
Procedural nausea (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 5 (6) | 7 (31)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 4 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 2 (2) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Cohort 2 (Limitation): Stimulated C-peptide data from the MMTT at Baseline and Week 26 showed undetectable C-peptide (<0.1 ng/mL) for all but one subject. For those subjects, AUC were not generated and assumed "zero" as serial undetectable C-peptide results cannot create a curve.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT04678557/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT04678557/SAP_001.pdf